CLINICAL TRIAL: NCT02627781
Title: Evaluation of Diagnostic Algorithm for Suspected Acute Appendicitis
Brief Title: Diagnostic Algorithm for Appendizitis (DIALAPP)
Acronym: DIALAPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Dr. Juliane Liese, MD, Goethe University
Other Study IDs: 268/15
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Reduction of Negative Appendectomy Rate
Keywords: acute appendicitis; Alvarado Score; negative appendectomy; right abdominal pain
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- suspected appendicitis: This group includes all patients with suspected appendicitis, who are admitted to our University Hospital.

SUMMARY:
The diagnosis of acute appendicitis remains a challenge in daily clinical practice. The high incidence of appendicitis drives the need to reduce morbidity and unnecessary costs due to negative appendectomies. The aim of the present observation study is to evaluate a diagnostic and therapeutic algorithm for suspected acute appendicitis.

The investigators believe that this diagnostic algorithm helps to simultaneously avoid unnecessary operations, costs and radiation exposure.

DETAILED DESCRIPTION:
This prospective observation study will be performed in the university hospital Frankfurt with a 24-h emergency service, with surgery and radiology readily available. The data will be compiled on patients older than 18 years who will be admitted to the emergency unit with suspected appendicitis.

During the study period, the clinical workflow is standardized. In all cases a resident of surgery and/or consultant surgeon clinically evaluate and perform an ultrasound scan on all patients with suspected appendicitis. With the use of clinical and laboratory results the physician (surgeon) will calculate the Alvarado Score and depending on the result the next diagnostic steps or the treatment will be chosen. Additionally, the department of gynecology of the university hospital routinely evaluate all women of childbearing age. Upon other terms following variables will be collected: age, gender, white blood cells (WBC), C-reactive protein (CRP), Alvarado Score, visuell pain scale, CT scan results, pathologic findings, time between admission and operation, operation procedure, treatment and diagnosis of patients without operation, length of hospital stay, and 30-day complication rate. Furthermore, there will be a follow-up of all patients (with and without operation) after 30 days and 6 months.

The investigators assume that the use of a diagnostic and therapeutic algorithm reduces unnecessary negative appendectomies and optimizes the duration of the hospital stay and the costs.

ELIGIBILITY:
Inclusion Criteria:

* complete evaluation, examination and diagnostic pathways of the patients with suspected appendicitis in our University Hospital

Exclusion Criteria:

* appendectomy during other operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our University department with suspected appendicitis and/or lower right abdominal pain.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the negative appendectomy rate | 6 months
  In this part of the study, the negative appendectomy rate will be determined. A negative appendectomy is characterized by normal findings in the pathological examination and therefore constitutes a medically unnecessary appendectomy.

SECONDARY OUTCOMES:
The influence of computed tomography for the diagnosis of acute appendicitis | 30 days
  In this part of the study the investigators evaluate the careful and cost-effective integration of computed tomography in the clinical pathway.
Incidence of readmission to hospital | 6 months
  In this part of the study the readmission rate to hospital will be evaluated because of postoperative complications, infections and continuous abdominal pain will be included.
Evaluation of postoperative complications | 6 months
  In all patients, who received an appendectomy the postoperative complication rate will be recorded. In statistical analysis factors, which are associated with complications will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Liese, MD, Principal Investigator — General and Visceral Surgery
Locations (1):
- Goethe University, Frankfurt, Germany

REFERENCES:
- [Derived] Malkomes P, Edmaier F, Liese J, Reinisch-Liese A, El Youzouri H, Schreckenbach T, Bucher AM, Bechstein WO, Schnitzbauer AA. DIALAPP: a prospective validation of a new diagnostic algorithm for acute appendicitis. Langenbecks Arch Surg. 2021 Feb;406(1):141-152. doi: 10.1007/s00423-020-02022-7. Epub 2020 Nov 19. PMID 33210209